CLINICAL TRIAL: NCT00684996
Title: A Phase I and a Randomized Phase II Study of Maximal Angiogenic Blockade in Advanced Renal Carcinoma: Bevacizumab (NSC-704865) With or Without MEDI-522 (NSC-719850)
Brief Title: Bevacizumab With or Without MEDI-522 in Treating Patients With Unresectable or Metastatic Kidney Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01099; NCI-2009-01099 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000596555; S0717 (Other: SWOG); S0717 (Other: CTEP); U10CA032102 (NIH)
Record Dates: First submitted 2008-05-24; First posted 2008-05-28 (Estimated); Results first posted 2014-01-14 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2013-04

CONDITIONS: Recurrent Renal Cell Cancer; Renal Cell Carcinoma; Stage III Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — etaracizumab; Bevacizumab

ARMS (2):
- Phase II Arm I (Active Comparator): Patients receive bevacizumab (10mg/kg) IV over 30-90 minutes on days 1 and 15.
  Interventions: Biological: bevacizumab
- Phase II Arm II (Active Comparator): Patients receive bevacizumab IV as in arm I at the RPTD determined in phase I, and humanized monoclonal antibody MEDI-522 (8mg/kg) IV over 30 minutes on days 1, 8, 15, and 22.
  Interventions: Drug: etaracizumab; Biological: bevacizumab

INTERVENTIONS:
Drug: etaracizumab — Given IV
  Other Names: Abegrin; humanized monoclonal antibody MEDI-522; MEDI-522; monoclonal antibody anti-alpha V beta 3 integrin MEDI-522
  Arms: Phase II Arm II
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF

SUMMARY:
This phase I/randomized phase II trial is studying the side effects and best dose of bevacizumab and to see how well it works when given together with or without MEDI-522 in treating patients with unresectable or metastatic kidney cancer. Monoclonal antibodies, such as bevacizumab and MEDI-522, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab and MEDI-522 may also stop the growth of tumor cells by blocking blood flow to the tumor. It is not yet known whether bevacizumab is more effective when given together with or without MEDI-522 in treating kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the appropriate dose of bevacizumab when administered with humanized monoclonal antibody MEDI-522 in patients with unresectable or metastatic renal cell carcinoma previously treated with sunitinib malate or sorafenib tosylate. (Phase I) II. To compare the progression-free survival of these patients treated with bevacizumab with versus without humanized monoclonal antibody MEDI-522. (Phase II) III. To evaluate the qualitative and quantitative toxicities of bevacizumab and humanized monoclonal antibody MEDI-522 in these patients. (Phase II) IV. To estimate overall survival and RECIST response rate (i.e., confirmed and unconfirmed, complete and partial responses) in both treatment arms. (Phase II)

OUTLINE: This is a multicenter, phase I, dose-escalation study of bevacizumab followed by a randomized phase II study.

PHASE I: Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and humanized monoclonal antibody MEDI-522 IV on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity until the recommended phase II dose (RPTD) of bevacizumab is determined.

PHASE II: Patients are stratified according to the number of prior treatment regimens for renal cell carcinoma (1 vs 2) and whether there is a clear cell component (yes vs no). Patients are randomized to 1 of 2 treatment arms:

ARM I: Patients receive bevacizumab (10 mg/kg) IV over 30-90 minutes on days 1 and 15.

ARM II: Patients receive bevacizumab IV as in arm I at the RPTD determined in phase I, and humanized monoclonal antibody MEDI-522 (8 mg/kg) IV over 30 minutes on days 1, 8, 15, and 22.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically for up to 3 years.

ELIGIBILITY:
Criteria:

* Histologically or cytologically confirmed renal cell carcinoma
* Metastatic or unresectable disease
* Must have received prior sunitinib malate or sorafenib tosylate for metastatic or unresectable disease
* Measurable disease
* No soft tissue disease that has been irradiated within the past 2 months
* More than 6 months since prior and no concurrent treated or untreated brain metastases
* Stable, treated brain metastases allowed provided they remained stable for more than 6 months
* Patients with clinical evidence of brain metastases must have a negative brain CT or MRI scan for metastatic disease
* Zubrod performance status 0-1
* Urine protein:creatinine ratio =< 0.5 OR urine protein < 1,000 mg by 24-hour collection
* Not be pregnant or nursing
* Fertile patients must use effective contraception during and for at least 6 months after completion of study therapy
* No serious or non-healing wound, ulcer, or bone fracture
* No clinically relevant bleeding diathesis or coagulopathy
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* No significant traumatic injury within the past 28 days
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No other prior malignancy, except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years
* No New York Heart Association class II-IV congestive heart failure
* No unstable symptomatic arrhythmia requiring medication
* Chronic, controlled arrhythmias (e.g., atrial fibrillation or paroxysmal supraventricular tachycardia) allowed
* None of the following cardiovascular conditions within the past 6 months: Arterial thrombosis, Unstable angina, Myocardial infarction, Cerebrovascular accident
* Must have controlled blood pressure, defined as systolic blood pressure (BP) =< 160 mm Hg and/or diastolic BP =< 90 mm Hg
* More than 7 days since prior core biopsy
* At least 14 days since completion of prior therapy and recovered
* At least 28 days since prior radiotherapy and recovered
* No prior radiotherapy to >= 25% of bone marrow
* No more than two prior systemic regimens for renal cell carcinoma (including adjuvant treatment)
* No prior bevacizumab or humanized monoclonal antibody MEDI-522
* No major surgical procedure or open biopsy within the past 28 days
* No concurrent need for a major surgical procedure
* Concurrent full-dose anticoagulation with warfarin allowed provided INR is between 2-3
* Concurrent low molecular weight heparin allowed
* No clinically significant vascular disease (e.g., aortic aneurysm or history of aortic dissection)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ryan, Principal Investigator — SWOG Cancer Research Network
Locations (5):
- United States (5):
  - Fremont - Rideout Cancer Center, Marysville, California
  - University of California at Davis Cancer Center, Sacramento, California
  - University of Michigan, Ann Arbor, Michigan
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - SWOG, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Bevacizumab (10 mg/kg) + MEDI-522: Patients receive bevacizumab (10/mg/kg or 5 mg/kg) IV over 30-90 minutes on days 1 and 15 and humanized monoclonal antibody MEDI-522 IV on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity until the recommended phase II dose (RPTD) of bevacizumab is determined.
Period: Overall Study
Arm/Group | Phase I Bevacizumab (10 mg/kg) + MEDI-522
Started | 5
Eligible | 5
Completed | 0
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Refusal unrelated to adverse event | 1
Not completed — Progression/relapse | 2
Not completed — Other reasons not protocol specified | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase I Bevacizumab (10 mg/kg) + MEDI-522: Patients receive bevacizumab (10 mg/kg or 5mg/kg) IV over 30-90 minutes on days 1 and 15 and humanized monoclonal antibody MEDI-522 IV on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity until the recommended phase II dose (RPTD) of bevacizumab is determined.
Arm/Group | Phase I Bevacizumab (10 mg/kg) + MEDI-522
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 61.5 [45.3 to 80.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Bevacizumab , Based on Incidence of Dose-limiting Toxicity (DLT) Graded According to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 (Phase I)
Time Frame: Up to 8 weeks
Population: The study was permanently closed to accrual on April 1, 2009, due to drug supply issues.
Groups:
- Phase I Bevacizumab (10 mg/kg) + MEDI-522: Patients receive bevacizumab (10 mg/kg or 5 mg/kg) IV over 30-90 minutes on days 1 and 15 and humanized monoclonal antibody MEDI-522 IV on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity until the recommended phase II dose (RPTD) of bevacizumab is determined.
Arm/Group | Phase I Bevacizumab (10 mg/kg) + MEDI-522
Number analyzed (Participants) | 0

2. Primary Outcome: Progression-free Survival (Phase II)
Description: Measured from date of registration to date of first observation of progressive disease, symptomatic deterioration or death due to any cause. Patients last known to be alive and progression-free are censored at date of last contact.
Time Frame: From date of registration to date of first observation of progressive disease, systemic deterioration, or death due to any cause, assessed up to 3 years
Population: The study was permanently closed to accrual on April 1, 2009, due to drug supply issues.
Arm/Group | Phase II Arm I | Phase II Arm II
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug, Graded According to NCI CTCAE Version 3.0 (Phase II)
Description: Adverse Events (AEs) are reported by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: Up to 3 years
Population: The study was permanently closed to accrual on April 1, 2009, due to drug supply issues.
Arm/Group | Phase II Arm I | Phase II Arm II
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Overall Survival (Phase II)
Description: Measure from date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: From date of registration to date of death due to any cause, assessed up to 3 years
Population: The study was permanently closed to accrual on April 1, 2009, due to drug supply issues.
Arm/Group | Phase II Arm I | Phase II Arm II
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Response Rate According to Response Evaluation Criteria in Solid Tumors (RECIST), Including Confirmed and Unconfirmed Complete and Partial Responses (Phase II)
Description: Complete Response (CR) is a complete disappearance of all measurable and non-measurable disease. No new lesions. No disease related symptoms. Partial Response (PR) applies only to patients with at least one measurable lesion. Greater than or equal to 30% decrease under baseline of the sum of longest diameters of all target measurable lesions. No unequivocal progression of nonmeasurable disease. No new lesions.
Time Frame: Up to 3 years
Population: The study was permanently closed to accrual on April 1, 2009, due to drug supply issues.
Arm/Group | Phase II Arm I | Phase II Arm II
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: as for outcome 3
Time Frame: Patients were assessed for the first 8 weeks for dose-limiting toxicities, then assessed for adverse events after every cycle (1 cycle = 28 days) of protocol treatment, up to 3 years
Population: Eligible patients who had received any treatment were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Groups:
- Phase I Bevacizumab (10 mg/kg) + MEDI-522: Patients receive bevacizumab (10/mg/kg or 5 mg/kg) IV over 30-90 minutes on days 1 and 15 and humanized monoclonal antibody MEDI-522 IV on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity un til the recommended phase II dose (RPTD) of bevacizumab is determined.
Arm/Group | Phase I Bevacizumab (10 mg/kg) + MEDI-522
Number analyzed (Participants) | 3
Participants
  Allergic reaction/hypersensitivity | 1
  Dyspnea (shortness of breath) | 1

ADVERSE EVENTS:
Time Frame: Patients were assessed for the first 8 weeks for dose-limiting toxicities, then assessed for adverse events after every cycle (1 cycle = 28 days) of protocol treatment, up to 3 years
Arm/Group | Phase I Bevacizumab (10 mg/kg) + MEDI-522
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Bevacizumab (10 mg/kg) + MEDI-522 (N=3)
Rigors/chills (General disorders) | 1
Allergic reaction/hypersensitivity (Immune system disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Bevacizumab (10 mg/kg) + MEDI-522 (N=3)
Hemoglobin (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pain - Esophagus (Gastrointestinal disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 2
Flu-like syndrome (General disorders) | 1
Rigors/chills (General disorders) | 2
Infection with unknown ANC - Upper airway NOS (Infections and infestations) | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1
AST, SGOT (Investigations) | 1
Alkaline phosphatase (Investigations) | 1
Creatinine (Investigations) | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1
Glomerular filtration rate (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less